CLINICAL TRIAL: NCT01847352
Title: Effect of Endogenous Iron Status on Hypoxic Pulmonary Vascular Responses and Their Attenuation by Intravenous Iron
Brief Title: Iron Status and Hypoxic Pulmonary Vascular Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 12/SC/0710
Record Dates: First submitted 2013-05-01; First posted 2013-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Lung Hypoxia; Pulmonary Arterial Hypertension; Iron Deficiency
Keywords: Hypoxia; Pulmonary hypertension; Iron deficiency; Hypoxic pulmonary vasoconstriction
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Iron Deficiencies; Hypoxia; Hypertension, Pulmonary | interventions — ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron-deficient (Other): Healthy volunteers meeting iron-deficient entry criteria; Intravenous administration of ferric carboxymaltose; Subacute hypoxic exposures
  Interventions: Drug: Intravenous administration of ferric carboxymaltose; Other: Subacute hypoxic exposures
- Iron-replete (Other): Healthy volunteers meeting iron-replete entry criteria; Intravenous administration of ferric carboxymaltose; Subacute hypoxic exposures
  Interventions: Drug: Intravenous administration of ferric carboxymaltose; Other: Subacute hypoxic exposures

INTERVENTIONS:
Drug: Intravenous administration of ferric carboxymaltose — Intravenous administration of ferric carboxymaltose 15mg/kg up to a maximum dose of 1000mg
  Other Names: Ferinject
Other: Subacute hypoxic exposures — Exposure to six hours of isocapnic hypoxia with end-tidal partial pressure of oxygen clamped at 55 Torr, with and without prior iron infusion
  Other Names: Hypoxia; Hypoxic challenge

SUMMARY:
On exposure to hypoxia (low oxygen) the normal response is for pulmonary arterial systolic blood pressure (PASP, blood pressure through the lungs) to increase. We have previously shown that raising iron by giving an infusion of iron into a vein reduces this pressure rise and that lowering iron by giving a drug that binds iron, magnifies this response. This is potentially a clinically important observation since iron-deficient people may be at increased risk of pulmonary hypertension if exposed transiently or permanently to hypoxia due to lung disease or residence at high altitude; furthermore if this were true then intravenous iron could be an important treatment in this patient group in the event of hypoxic exposure. The observed effects of iron on PASP are likely to be because iron levels affect oxygen sensing. Low iron levels make the body behave as if exposed to low oxygen by inhibiting the breakdown of the family of oxygen-sensing transcription factors, 'hypoxia inducible factor' or HIF. This includes one of the body's normal responses to low oxygen levels - raising blood pressure through the lungs.

This study will answer the question (1) do iron-deficient volunteers have a greater rise in PASP with hypoxia than those who are iron-replete, and (2) does giving intravenous iron cause a greater reduction in the rise in PASP in those who are iron-deficient than iron-replete? The purpose of this study is not to test the safety or clinical efficacy of iron which is already known.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study
* Men and women aged 18 years or older and generally in good health
* Detectable tricuspid regurgitation on echocardiography during both normoxia and hypoxia enabling measurement of pulmonary arterial pressure
* For iron-deficient volunteers: ferritin ≤15microg/L and transferrin saturation <16%
* For iron-replete volunteers: ferritin ≥20microg/L and transferrin saturation ≥20%

Exclusion Criteria:

* Haemoglobin <8.0g/dl
* Haemoglobinopathy
* Iron overload defined as ferritin >300microg/L
* Hypoxia at rest or on walking (SaO2 <94%) or significant comorbidity that may affect haematinics, pulmonary vascular or ventilatory responses, e.g. current infection, a chronic inflammatory condition, known cardiovalvular lesion or pulmonary hypertension, uncontrolled asthma or chronic obstructive pulmonary disease
* Exposure to high altitude (>2,500m) within the previous six weeks or air travel >4 hours within the previous week
* Iron supplementation or blood transfusion within the previous 6 weeks
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
∆PASP in iron-replete compared to iron-deficient volunteers | During six hours of hypoxia without prior iron infusion
  Difference between the rise in pulmonary artery systolic pressure during a hypoxic challenge in iron-replete compared to iron-deficient volunteers

SECONDARY OUTCOMES:
∆PASP, with versus without prior iron infusion, in iron-replete compared to iron-deficient volunteers | During two six-hour periods of hypoxia; assessments separated by at least a week
  Difference between the rise in pulmonary artery systolic pressure during a hypoxic challenge in iron-replete compared to iron-deficient volunteers, with versus without a prior iron infusion
Blood parameter changes, pre- versus post-intravenous iron, in iron-replete compared to iron-deficient volunteers | After six hours of hypoxia, at both study assessments
Ventilation parameter changes, pre- versus post-intravenous iron, in iron-replete compared to iron-deficient volunteers | During six hours of hypoxia, at both study assessments

OTHER OUTCOMES:
Fatigue scores in iron-replete versus iron-deficient volunteers | Assessed at baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Annabel H Nickol, MBBS PhD, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford Department of Physiology, Anatomy and Genetics, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith TG, Balanos GM, Croft QP, Talbot NP, Dorrington KL, Ratcliffe PJ, Robbins PA. The increase in pulmonary arterial pressure caused by hypoxia depends on iron status. J Physiol. 2008 Dec 15;586(24):5999-6005. doi: 10.1113/jphysiol.2008.160960. Epub 2008 Oct 27. PMID 18955380
- [Background] Smith TG, Talbot NP, Privat C, Rivera-Ch M, Nickol AH, Ratcliffe PJ, Dorrington KL, Leon-Velarde F, Robbins PA. Effects of iron supplementation and depletion on hypoxic pulmonary hypertension: two randomized controlled trials. JAMA. 2009 Oct 7;302(13):1444-50. doi: 10.1001/jama.2009.1404. PMID 19809026
- [Background] Talbot NP, Smith TG, Privat C, Nickol AH, Rivera-Ch M, Leon-Velarde F, Dorrington KL, Robbins PA. Intravenous iron supplementation may protect against acute mountain sickness: a randomized, double-blinded, placebo-controlled trial. High Alt Med Biol. 2011 Fall;12(3):265-9. doi: 10.1089/ham.2011.1005. PMID 21962070
- [Background] Balanos GM, Dorrington KL, Robbins PA. Desferrioxamine elevates pulmonary vascular resistance in humans: potential for involvement of HIF-1. J Appl Physiol (1985). 2002 Jun;92(6):2501-7. doi: 10.1152/japplphysiol.00965.2001. PMID 12015365
- [Result] Frise MC, Cheng HY, Nickol AH, Curtis MK, Pollard KA, Roberts DJ, Ratcliffe PJ, Dorrington KL, Robbins PA. Clinical iron deficiency disturbs normal human responses to hypoxia. J Clin Invest. 2016 Jun 1;126(6):2139-50. doi: 10.1172/JCI85715. Epub 2016 May 3. PMID 27140401
- See also: Research Group Website — http://www.dpag.ox.ac.uk/team/peter-robbins
- See also: Funding Body Website — https://www.bhf.org.uk/research-projects/effects-of-iron-deficiency-and-intravenous-iron-on-human-cardiorespiratory-physiology